CLINICAL TRIAL: NCT03025659
Title: Characterization of Lactic Acidosis in Pediatric Postoperative Cardiac Patients
Brief Title: Lactate Acidosis in Postoperative Hearts
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201601991
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Post-cardiac Surgery; Hyperlactatemia
Keywords: pediatric; congenital heart disease
MeSH Terms: conditions — Hyperlactatemia; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric post-cardiac surgery: All immediately post-operative pediatric cardiac patients will be enrolled. Standard of care laboratory analysis will be performed based on current clinical protocols. Results for lactate, blood gases, liver enzymes, creatinine, glucose, hemoglobin, hematocrit and other direct and indirect measure of cardiac output will be collected. Investigators will also measure pyruvate levels at specific time points, which is not part of standard of care. To measure pyruvate, an additional 1 ml of arterial blood will be drawn at each routine postoperative blood draw. The lactate/pyruvate ratio will be calculated and compared to direct and indirect measure of cardiac output described above.
  Interventions: Other: Pyruvate levels

INTERVENTIONS:
Other: Pyruvate levels — An additional 1 ml of arterial blood will be drawn at each routine postoperative blood draw (Hour 0, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 for participants 10kg and above or only at Hour 0, 2, 4, 6, 8, and 12 for infants under 10 kg) to measure the concentration of pyruvate in blood.

SUMMARY:
This is a single-center, observational study. Investigators aim to characterize the metabolism of lactate in children over the first forty-eight hours following cardiac surgery. Blood samples will be obtained up to 12 timepoints. Samples will be analyzed for concentration of pyruvate. Results will be compared to standard of care laboratory results for lactate and other direct and indirect measures of cardiac output.

DETAILED DESCRIPTION:
Investigators will characterize the etiologies of hyperlactatemia predominantly present at serial postoperative timepoints in children recovering from cardiac surgery by following lactate levels and the lactate-to-pyruvate ratio over the first 48 post-operative hours and correlating them with cardiac output as determined by conventional markers and physical exam. Investigators expect to validate the assumption that in children recovering from heart surgery whose cardiac output is apparently normal, hyperlactatemia (if seen) is predominantly due to impaired lactate clearance or metabolism, while in those whose cardiac output is low, it is predominantly due to inadequate oxygen delivery. Blood samples will be obtained up to 12 timepoints (arrival at the intensive care unit postoperatively, hour 1, hour 2, hour 3, hour 4, hour 6, hour 8, hour 10, hour 12, hour 24, hour 36 and hour 48 postoperative) or only at up to 6 time points (approximately Hour 0, 2, 4, 6, 8, and 12) for infants under 10 kg as described below. . Samples will be analyzed for concentration of pyruvate. Results will be compared to standard of care laboratory results for lactate and other direct and indirect measures of cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* All immediately post-operative cardiac patients admitted to the pediatric cardiac intensive care unit (PCICU)

Exclusion Criteria:

* Lack of parental or patient consent, or patient assent when applicable, including non-English speakers and wards of the state
* Dosing weight less than 4 kg*
* Cardiac catheterization being the only operative procedure
* Severe hepatic dysfunction at any time during the hospital course
* Seizures during the study period
* Sepsis during the study period
* Need for extracorporeal membrane oxygenation or continuous renal replacement therapy
* Known congenital myopathy, ataxia, polyneuropathies or inborn errors of metabolism including congenital lactic acidosis and other mitochondrial disorders
* Primary hypoventilation
* Malignancies
* Fanconi syndrome
* Wernicke encephalopathy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cardiac surgical patients at UF Health Shands Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-05-28 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Lactate/pyruvate ratio | Hourly, assessed up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Tsifansky, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Shands Children's Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected on REDCap (secure web application for building and managing online surveys and databases) and available to study staff via password protected access